CLINICAL TRIAL: NCT02847572
Title: A Clinical Assessment of Visual Performance of Combining the Tecnis Symfony Extended Range of Vision IOL (ZXR00) With the +3.25D Tecnis Multifocal 1-Piece IOL (ZLB00) in Subjects Undergoing Bilateral Cataract Extraction
Brief Title: Assessment of Visual Performance Combining a Symfony IOL and a +3.25 Tecnis Multifocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crystal Clear Vision (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CrystalClearVision
Record Dates: First submitted 2016-03-01; First posted 2016-07-28 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery Patient (Other): All patients to be implanted bilaterally with a Tecnis Extended Range Lens in the Dominant eye and a Low Add Multifocal in the non dominant
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Procedure: Cataract Surgery — All patients wil be having intraocular lens surgery

SUMMARY:
This will be a single center, non comparison clinical trial. Fifty study patients will have the Symfony IOL implanted in their dominant eye and a +3,25D Tecnis Multifocal in their non-dominant eye. The investigators will be evaluated vision at distance, intermediate and near as well as assessing patient satisfaction and spectacle independence.

DETAILED DESCRIPTION:
Each study patient will undergo the same routine cataract extraction procedure in each eye. In their dominant eye a Tecnis Symfony IOL will be implanted and in the non dominant eye, a Tecnis +3.25D Multifocal implanted. The surgeries will be within 2 days of each other. Every patient will receive same postoperative instructions and medications. The aim is to investigate the potential benefits of implanting two different IOL's to give the patient a wider range of near vision with decreased risk of haloing and glare to enable them to be less dependent on reading glasses

ELIGIBILITY:
Inclusion Criteria:

* good general health,
* willing to comply with study instructions,
* Visual potential of 20/30 or better,
* less than 1.5D of corneal astigmatism,
* normal macula,
* clear lens or cataract,
* pupil size greater than 3.5mm

Exclusion Criteria:

* known pathology to affect visual outcome,
* amblyopia or strabismus,
* pupil abnormalities,
* zonule problems,
* keratoconus,
* no prior ocular surgery,use of medication that could affect vision,
* uncontrolled systemic disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 months
  Vision will be measured at distance, intermediate and near with and without correction.

SECONDARY OUTCOMES:
Patient Satisfaction | 3 months
  Patients will fill in a Patient Satisfaction Questionnaire at all visits. Contrast sensitivity will also be measured

CONTACTS AND LOCATIONS:
Overall Officials: Sondra Black, OD, Study Chair — Crystal Clear Vision
Locations (1):
- Crystal Clear Vision, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No